CLINICAL TRIAL: NCT05930990
Title: Mamas in Harmony: a Feasibility Study With Pilot Randomised Controlled Trial and Process Evaluation of a Music and Social Support Group Intervention for Postnatal Mothers and Their Infants
Brief Title: Feasibility Study of a Music and Social Support Intervention for Postnatal Mothers/Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Responsible Party: Principal Investigator, Fiona Lynn, Principal Investigator, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MHLS 22_168
Record Dates: First submitted 2023-04-03; First posted 2023-07-05 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Anxiety
Keywords: Depression; Stress; Parenting confidence; Social support; Mother-infant attachment; Health related quality of life
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mamas in Harmony (and usual care) (Experimental): Mamas in Harmony is a 1 hour face to face intervention for mothers and their infants, delivered in groups of 10-12 mother-infant dyads, every week for 8 weeks. Mothers and infants also receive usual postnatal care from health and social care services.
  Interventions: Behavioral: Mamas in Harmony
- Control (usual care only) (No Intervention): Mothers and infants receive usual postnatal care from health and social care services.

INTERVENTIONS:
Behavioral: Mamas in Harmony — Mothers attend 8x 1 hour weekly classes with their infant. Classes take place in a community venue. Mothers sit with their infant on the floor in circle formation on cushioned mats. Group singing facilitated for 40 minutes by the intervention facilitator, a professional musician/choir leader. A mix of songs are introduced that are easy to learn without the need for lyric sheets. Mothers will be encouraged to sing along. Mothers will be encouraged to interact with their infant through various sensory stimuli involving touch, sound and visual. The end of each singing session involves a short period of quiet time, soothing sounds are provided by the intervention facilitator using voice and instruments. 20 minutes of facilitated social support will follow and mothers will be provided with refreshments. Mothers will be encouraged to interact with other mothers to promote social connection.
  Arms: Mamas in Harmony (and usual care)

SUMMARY:
This research study aims to assess the feasibility of conducting a full scale trial of Mamas in Harmony, a group music and social support class delivered by a professional musician for mothers and their babies. Classes for Mamas in Harmony run for 1 hour each week for 8 weeks at a community venue with 10-12 mothers and babies in each class.

The aim of this study is to conduct a pilot randomised controlled trial and process evaluation to assess recruitment rate, retention rate, adherence rate to the study protocol, attendance rate for the intervention, completion rate of outcome measurement tools, acceptability of the intervention, and barriers/facilitators for study participation and intervention delivery.

This feasibility study aims to recruit 60 mothers and babies. Forty will be randomly allocated to the intervention group of Mamas in Harmony and receive standard postnatal care and twenty will receive standard postnatal care only, as the control group.

All mothers will be asked to complete study questionnaires at three time points over a 6 month period to assess their mental health and wellbeing and bonding with their baby.

Mothers will also be asked if they wish to share their opinions and experiences about the research study and Mamas in Harmony classes (if they were allocated to that group) in an interview, to provide their thoughts, whether anything made it easy/difficult for them to participate and whether they have any suggestions on how to improve the study procedure.

The musician will also be asked for their experiences on the barriers and facilitators of intervention delivery.

DETAILED DESCRIPTION:
Perinatal mental health problems have the potential to lead to multiple negative outcomes for both mother and child, and mental health in the perinatal period is a current leading public health issue with significant economic burden if untreated. The perinatal period lasts for the duration of pregnancy and for 1 year after the birth of the child. Symptoms of low mood, anxiety, stress, feeling isolated, and difficulties with mother-infant attachment are frequently experienced by both antenatal and postnatal mothers. It is reported that anxiety is often overlooked in the perinatal period, with limited research carried out in relation to perinatal anxiety compared to depression, with little knowledge around epidemiology or effectiveness of interventions for perinatal mental health conditions other than postnatal depression (PND). This is despite associations found between maternal anxiety and adverse outcomes for the child.

Studies investigating the effect of poor postnatal mental health have found an adverse impact on mother-infant attachment, bonding, self-regulation and empathy. Consequently, mothers find it difficult to engage with their infants both emotionally and behaviourally resulting in reducing their physical contact.

Regular screening for perinatal depression and anxiety disorders by health professionals is recommended in the UK by National Institute for Health and Care Excellence (NICE) guidelines from the first contact with the mother, throughout pregnancy and the postnatal period using assessment tools. However, postnatal mental health problems often go unidentified, undiagnosed, and untreated for many women or they do not meet the eligibility threshold for specialist mental health services after the birth of their baby.

Current pharmacological treatment options offered by health professionals involved in the care of mothers often have potential for side effects and low uptake and adherence, especially for breastfeeding mothers. Psychotherapy has presented challenges of mixed results, and short-lived improvements. Consequently there has been an increase in interest in non-pharmacological interventions, such as arts in health programmes.

Strong evidence supports the arts in improving wellbeing and quality of life among adults. Arts in health activities are wide ranging and, in particular, include performing arts, such as music. The gap that remains in current literature is an arts in health based group intervention for mother-infant dyads, supporting the reduction in symptoms of anxiety and stress, promoting social support and targeting an improvement in the mother-infant relationship.

This study will seek to explore the feasibility and the potential benefit of a new mother-infant group intervention, Mamas in Harmony, that combines group music classes with social support using a pilot randomised controlled trial and process evaluation.

Sixty mother-infant dyads aim to be recruited via social media, including Facebook and Twitter, and recruitment posters on communal/public facing noticeboards. Local Women's and Community Centres, community mother and baby classes, social support organisations and SureStart Children's Centres (Department for Education funded) will be asked to display posters/flyers. Following informed consent and baseline data collection, mothers will be randomly allocated using a 2:1 ratio to the intervention or control group. Mamas in Harmony sessions will be delivered by a professional musician/choir leader in a community venue face to face in groups of 10-12 mother-infant dyads, for 1 hour each week for 8 weeks along with their usual postnatal care from health and social care services. The control group receive usual postnatal care only.

All mothers will be invited to complete questionnaires at baseline (prior to randomisation), 3 months and 6 months post-randomisation either online or posted in paper format to assess completion rates of measurement tools for anxiety, depression, perceived stress, parenting confidence, perceived social support, mother-infant attachment, health related quality of life and service and resource use.

Study registers will be used to assess recruitment rate, retention rate, adherence to the study protocol and attendance rate for the intervention.

Evaluation forms will be administered to the intervention group in week 8 and semi structured interviews completed online with a subset of 8 mothers from intervention and control groups at the end of the study to establish acceptability, and maternal satisfaction with the intervention and/or research study, as applicable. Semi structured interview/s will be conducted with the intervention facilitator/s to allow an understanding of the facilitators' perspectives of barriers and facilitators for intervention delivery.

ELIGIBILITY:
Inclusion Criteria:

* Mothers who have a baby aged ≥14 days to ≤4 months at time of consent.
* Able and willing to provide consent identified by having a satisfactory understanding of English and comprehension of the participant information sheet and consent form.

Exclusion Criteria:

* Mothers who have given birth in the last 14 days.
* Infants >4 months at time of consent.
* Identified as not having satisfactory understanding of English and comprehension of the participant information sheet and consent form.
* Mothers who have received a diagnosis of, or being treated for, severe mental illness including Bipolar disorder, Psychoses or Schizophrenia within the past 6 months (discovered through self-report at time of eligibility screening).

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Individuals who have given birth, who may not identify as women.
Enrollment: 72 (Actual)
Dates: Start 2023-03-16 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2024-04-12 (Actual)

PRIMARY OUTCOMES:
Rates of recruitment and retention | 6 months
  Rates of participant flow through each stage of the pilot RCT, from participant invite for eligibility assessment through to outcome assessment at 6-month follow-up, using screening logs and study registers. Data supplemented with reasons for non-participation, if disclosed.

SECONDARY OUTCOMES:
Rate of adherence to the study protocol | 6 months
  Rate of adherence of participants across each stage of the pilot RCT, using study registers. Data supplemented with reasons for non-participation, if disclosed.
Rate of attendance to Mamas in Harmony intervention sessions | 8 weeks
  Rate of attendance of participants allocated to the intervention group using study registers. Data supplemented with reasons for non-attendance, if disclosed.
Completion rate of the Generalised Anxiety Disorder-7 scale (GAD-7) | 3 months and 6 months post randomisation
  Developed to assist health professionals in detecting generalised anxiety. GAD-7 consists of 7 questions with a choice of 4 responses based on how the individual has felt over the past 2 weeks. Measured on a scale of 0-21. Scores of 5, 10 and 15 are taken as the cut off points for mild, moderate and severe anxiety respectively. When used as a screening tool, further evaluation is recommended when the score is 10 or greater. This scale will be administered to assess whether it is an appropriate outcome measure for a full scale trial, as determined by completion rate and proportion of missing data.
Completion rate of the Edinburgh Postnatal Depression Scale (EPDS) | 3 months and 6 months post randomisation
  Developed to assist health professionals in detecting postnatal depression. Scale consists of 10 questions with a choice of 4 responses based on how the individual has felt over the past 7 days. Measured on a scale of 0-30. A score of more than 10 suggests depression may be present and further evaluation is recommended. This scale will be administered to assess whether it is an appropriate outcome measure for a full scale trial, as determined by completion rate and proportion of missing data.
Completion rate of the Perceived Stress Scale (PSS) | 3 months and 6 months post randomisation
  Developed to assist in assessing stress level in young people and adults aged 12 and above. It evaluates the degree to which an individual has perceived life as unpredictable, uncontrollable and overloading over the previous month. Consisting of 10 questions. The PSS score is obtained by summing across all items. Higher scores indicate higher levels of perceived stress, There are no published score cut-offs as this is not a diagnostic instrument. This scale will be administered to assess whether it is an appropriate outcome measure for a full scale trial, as determined by completion rate and proportion of missing data.
Completion rate of the Karitane Parenting Confidence Scale (KPCS) | 3 months and 6 months post randomisation
  Developed to assist in the support and development of parenting skills for parents of children 0-12 months of age. Containing 15 items with scores of 0-45. Parents scoring 39 or less may be experiencing low levels of parenting confidence. This scale will be administered to assess whether it is an appropriate outcome measure for a full scale trial, as determined by completion rate and proportion of missing data.
Completion rate of the Social Support Survey (SSS) | 3 months and 6 months post randomisation
  Consisting of 19 questions across 4 separate social support subscales and an overall functional social support index. A higher score for an individual scale or for the overall support index indicates more support. This tool will be administered to assess whether it is an appropriate outcome measure for a full scale trial, as determined by completion rate and proportion of missing data.
Completion rate of the Maternal Postnatal Attachment Scale (MPAS) | 3 months and 6 months post randomisation
  Developed to assess the mothers emotional response to her infant along a number of dimensions relating to parent-infant attachment. 19 items and number of response categories varies between two and five. Item totals are summed to obtain the scale score. Lower scores indicate lower attachment and vice versa. This scale will be administered to assess whether it is an appropriate outcome measure for a full scale trial, as determined by completion rate and proportion of missing data.
Completion rate of the EuroQol EQ-5D-5L | 3 months and 6 months post randomisation
  Respondents rate their health-related quality of life today on 5 dimensions (mobility, self care, usual activities, pain/discomfort and anxiety/depression) in order to assess treatment effects and investigate gains (or losses) in reported health status. This tool will be administered to assess whether it is an appropriate outcome measure for a full scale trial, as determined by completion rate and proportion of missing data.
Completion rate of service and resource use log | 3 and 6 months
  A service and resource use instrument has been developed for use in this study to capture and cost public sector service and resource use for postnatal mothers. This will be administered to assess whether it is an appropriate outcome measure for a full scale trial, as determined by completion rate and proportion of missing data.
Satisfaction of Mamas in Harmony intervention | 8 weeks
  To explore expectations of and satisfaction with the intervention and ideas for improvement using evaluation forms administered to mothers in week 8 at the final session of the intervention, including a scale of 0-10, a higher score indicating a better rating, scale of strongly disagree to strongly agree, scale of very unlikely to very likely, multiple choice questions and free text answer boxes.
Acceptability of Mamas in Harmony intervention | 6 months
  Gain insight on the acceptability of the intervention in terms of being liked or disliked, appropriate, benefits gained, to identify any barriers to attendance and/or engagement that exist and recommendations for improvement using semi-structured interviews with a subset of participants
Perspectives on barriers and facilitators to intervention delivery | 6 months
  Understand perspectives on barriers and facilitators to intervention delivery to determine improvements needed for future research using a semi-structured interview with the intervention facilitator/s.
Perspectives on barriers and facilitators to study participation | 6 months
  Understand perspectives on barriers and facilitators to study participation using semi-structured interviews with a subgroup of study participants
Perspectives on intervention fidelity | 6 months
  Understand perspectives on implementation in terms of fidelity (intervention delivered as intended) using semi-structured interviews with intervention facilitators

CONTACTS AND LOCATIONS:
Overall Officials: Fiona A Lynn, PhD, Principal Investigator — Queen's University, Belfast
Locations (1):
- Queen's University, Belfast, County Antrim, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Colella CA, McNeill J, McCann U, Lynn FA. Mamas in Harmony: protocol for a pilot RCT and process evaluation of a music and social support intervention establishing the feasibility of reducing anxiety and stress in postnatal mothers. Pilot Feasibility Stud. 2025 Apr 10;11(1):44. doi: 10.1186/s40814-025-01629-1. PMID 40211322
- See also: Study webpage — http://go.qub.ac.uk/mamasinharmony

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2023-02-13): https://cdn.clinicaltrials.gov/large-docs/90/NCT05930990/Prot_ICF_000.pdf